CLINICAL TRIAL: NCT03764982
Title: RehabNytte - A Multi Center Study in Specialized Rehabilitation Centers in Norway Exploring Health, Function, Workability and Quality of Life Following Rehabilitation
Brief Title: RehabNytte - A Study of Rehabilitation Processes in Specialized Care in Norway
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: VIRKE Rehab (Unknown); Norwegian National Centre for Occupational Rehabilitation (NKARR) (Unknown); Regional Center of Knowledge Translation in Rehabilitation, Sunnaas rehabilitation hosp. (Unknown); Skogli Health and Rehabilitation Center (Other); Stiftelsen CatoSenteret rehabilitation center (Unknown); HLF Briskeby rehabilitation center (Unknown); Vikersund rehabilitation center and kurbad (Unknown); Røysumtunet rehabilitation center (Unknown); Evjeklinikken (Other); Montebellosenteret (Unknown); Muritunet as rehabilitation center (Unknown); Røde Kors Haugland rehabilitation center (Other); Sørlandet rehabilitation center (Unknown); AVONOVA Ringerike rehabilitation (Unknown); Hernes institute (Unknown); NKS Helsehus as (Unknown); Ravneberghaugen rehabilitation center (Unknown); Åstveit rehabilitation center (Unknown); Selli rehabilitation center (Unknown); Helsepartner rehabilitation center (Unknown); Norwegian National Advisory Unit on Rehabilitation in Rheumatology (NKRR) (Unknown); REMEDY - Center for treatment of Rheumatic and Musculoskeletal Diseases (Unknown)
Responsible Party: Principal Investigator, Rikke Helene Moe, Principal Investigator, Diakonhjemmet Hospital
Other Study IDs: 99008; DS-00040 (Registry Identifier: Data protection approval)
Record Dates: First submitted 2018-11-23; First posted 2018-12-05 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Rehabilitation
Keywords: Rehabilitation; Multidisciplinary; Health care; *the RehabNytte Consortium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study is to describe function and health related to quality of life during the first year after rehabilitation, to measure the degree and impact of user involvement in the rehabilitation process, assess factors associated with change in work -ability and -participation, and to test measurement properties of a new core set of outcome measures for rehabilitation launched by the Norwegian Directorate of Health.

DETAILED DESCRIPTION:
This is a large multicentre cohort study including patients receiving rehabilitation at 17 rehabilitation centres from Norway, *the RehabNytte Consortium. Invitation and registration of participants will be conducted by local project coordinators in the period between 01.01.2019 and 31.03.2020.

All participants will receive rehabilitation as usual at each centre, and report HRQoL, health and function (by PROMS) through a digital self-reporting system at admission, discharge and after 3, 6 and 12 months.

This study seeks to answer several research questions related to the overarching areas:

1. Patient reported change of function, health and quality of life during the first year after rehabilitation
2. Degree of user involvement in rehabilitation
3. Change in work -ability and -participation
4. Quality assessment (use of Quality indicator set)
5. Measurement characteristics (feasibility and responsiveness) of recommended PROMS in rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Patients that participates in inpatient or outpatient rehabilitation programs at one of the participating centers.
* Age over 18 years
* Access to internet at home
* Access to personal secure login with BANK ID.

Exclusion Criteria:

* Severely reduced cognitive function
* severe mental illness with inadequate consent competence ability to participate
* Insufficient understanding of Norwegian written language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients receiving rehabilitation at seventeen rehabilitation centres in specialist care (all health regions)
  * All diagnoses, with largest groups of musculoskeletal diseases, neurological conditions (stroke, MS), cancer, and heart- and lunge conditions.
Sampling Method: Non-Probability Sample
Enrollment: 3793 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The EuroQoL-5D-5L | 1-3 minutes
  5-item questionnaire assessing function and health in walking, ADL, personal care, pain/discomfort and anxiety/depression. Sores could be calculated both as numbers and 'utilities'.
The EuroQoL-VAS health | 1-2 minutes
  The EUROQUOL 5D-5L includes a 100 mm VAS scale/thermometer. Index value: 0-1, 1 is best VAS gen health: 0-100, 100 is best
The Patient Specific Functional Scale (PSFS) | 2-6 minutes
  Patient-specific instrument. Up to five activities are described by the patient, and scored according to experienced performance (0-10, 10 is best).
PROMIS 29 | 5-10 minutes
  The PROMIS-29, a generic health-related quality of life survey, assesses each of the 7 PROMIS domains (depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities) with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity.

OTHER OUTCOMES:
The MUSS Quality Indicator set for Rehabilitation | 3-8 minutes
  This Quality Indicator assessment tool consist of two separate questionnaires answered by rehabilitation managers and patients, and each questionnaire consist of 10 and 11 questions respectively. The quality indicators are originally developed for use in Rheumatic and musculoskeletal disorders (RMDs) has been developed and pilot tested according to the Rand/UCLA Appropriateness Method. In this study the set will be tested in a generic population.

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, Professor, Study Director — Dep.Rheumatology, Diakonhjemmet hospital
Locations (17):
- Norway (17):
  - Helsepartner rehabilitation centre, Alta
  - Åstveit rehabilitation centre, Bergen
  - Sørlandet rehabilitation centre, Eiken
  - Evjeklinikken rehabilitation centre, Evje
  - Red Cross Haugland rehabilitation centre, Flekke
  - Ravneberghaugen rehabilitation centre, Hagavik
  - Hernes institutt, Hernes
  - AVONOVA Ringerike rehabilitation centre, Hønefoss
  - Røysumtunet rehabiliteringssenter, Jaren
  - Selli rehabilitation centre, Klæbu
  - HLF Briskeby rehabilitation centre, Lier
  - Montebellosenteret, Lillehammer
  - Skogli rehabilitation centre, Lillehammer
  - NKS Helsehus, Lørenskog
  - CatoSenteret, Son
  - Muritunet rehabilitation centre, Valldal
  - Vikersund rehabilitation centre, Vikersund

IPD SHARING:
Plan to Share IPD: Undecided
Participating centres will have access to de-identificated IPD after the data collection period is completed. Data will only be shared with other researchers after approval by the steering committee, and in line with the purposes of the project.

REFERENCES:
- [Derived] Skinnes MN, Uhlig T, Johansen T, Morvik HK, Farsund N, Fossen J, Skardal RF, Tollin G, Degirmenci AET, Habberstad A, Sexton J, Kollerud R, Kjeken I; RehabNytte Consortium; Wilkie R, Moe RH. Exploring differences in health-related benefit status in the year before, during and after specialist rehabilitation: a Norwegian case-control study. BMJ Open. 2026 Jan 21;16(1):e105722. doi: 10.1136/bmjopen-2025-105722. PMID 41565335
- [Derived] Rimehaug SA, Moe RH, Dagfinrud H, Fischer F, Johansen T, Kjeken I, Klokkerud M, Fossmo HL, Lyken AD, Kvalheim TR, Soldal S, Sand-Svartrud AL; RehabNytte Consortium. Measurement properties of the PROMIS-29 profile v2.1 in a Norwegian rehabilitation context. J Patient Rep Outcomes. 2025 Jul 31;9(1):98. doi: 10.1186/s41687-025-00929-7. PMID 40742502
- [Derived] Sand-Svartrud AL, Dagfinrud H, Fossen J, Framstad H, Irgens EL, Morvik HK, Sexton J, Moe RH, Kjeken I. Impact of provider feedback on quality improvement in rehabilitation services: an interrupted time series analysis. Front Rehabil Sci. 2025 Mar 6;6:1564346. doi: 10.3389/fresc.2025.1564346. eCollection 2025. PMID 40115421
- [Derived] Sand-Svartrud AL, Kjeken I, Skardal RF, Gjerset GM, Johnsen TJ, Lyken AD, Dagfinrud H, Moe RH. Completeness of repeated patient-reported outcome measures in adult rehabilitation: a randomized controlled trial in a diverse clinical population. BMC Health Serv Res. 2024 Dec 24;24(1):1648. doi: 10.1186/s12913-024-12103-8. PMID 39716127